CLINICAL TRIAL: NCT03102424
Title: A Prospective, Double Blind, Randomized, Placebo- Controlled Trial of Transcutaneous Electrical Nerve Stimulator (DW1330) to Improve Blood Glucose Control in Patients With Type 2 Diabetes
Brief Title: Transcutaneous Electrical Nerve Stimulator to Improve Blood Glucose Control in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiwan Resonant Waves Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TRWRDM1604001; 1056030994 (Other Grant/Funding Number: Taiwan: Food and Drugs Administration (TFDA))
Record Dates: First submitted 2016-12-26; First posted 2017-04-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Nerve Stimulator (DW1330) (Experimental): The 20 weeks of treatment of the DW1330 device, all the patients enrolled should perform 1 treatment within 1 hour after dinner 5 days a week.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulator (DW1330)
- Sham DW1330 device (Placebo Comparator): The 20 weeks of treatment of the Sham DW1330 device, all the patients enrolled should perform 1 treatment within 1 hour after dinner 5 days a week.
  Interventions: Device: Sham DW1330 device

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulator (DW1330) — The 20 weeks of treatment of the DW1330 device, all the patients enrolled should perform 1 treatment within 1 hour after dinner 5 days a week.
  Other Names: Dragon Waves Resonant Home Care Electronic Nerve Stimulator (DW1330); DW1330; T2DM-MENS
  Arms: Transcutaneous Electrical Nerve Stimulator (DW1330)
Device: Sham DW1330 device — The Sham DW1330 device will be masked by the same appearance as the study device (DW1330). The usage of time and location of Sham DW1330 device will be completely the same with study device (DW1330). However, the electronic model, including the frequency and time consistence of electronic stimulation are different between the Sham DW1330 device and the study device (DW1330). The 20 weeks of treatment of the DW1330 device, all the patients enrolled should perform 1 treatment within 1 hour after dinner 5 days a week.
  Arms: Sham DW1330 device

SUMMARY:
The primary study objective is to demonstrate the use of "Dragon Waves Resonant Home Care" Electronic Nerve Stimulator (DW1330) is associated with improvement of blood glucose control, as measured by change of glycated hemoglobin (HbA1c). The second study objectives are to demonstrate that DW1330 is associated with the mechanism of glycemic control and inflammation pathways. The study is also aimed to investigate the safety of DW1330.

DETAILED DESCRIPTION:
This is a multi-center, prospective, double blind, randomized, placebo-controlled trial of transcutaneous electrical nerve stimulator (DW1330) to improve blood glucose control in patients with type 2 diabetes. Subjects with type 2 diabetes who meet inclusion/exclusion criteria will be randomized to either of the 2 groups below:

1. DW1330
2. Placebo (sham TENS delivering ineffective pulse wave)

After enrollment, subjects will be randomly assigned to receive one of the study treatments in a double-blind fashion. All patients enrolled should perform 1 treatment within 1 hour after dinner 5 days a week. The end of a 20 week treatment period, subjects will be followed for an additional 2 weeks for safety follow-up. The time frame includes 2 weeks of screening, 20 weeks of treatment, and 2 weeks of post-treatment follow-up.

Study visits will occur every 2 or 4 weeks depending on the study phase. At randomization visit study device will be dispensed at the site, during the treatment period visits, all Adverse Events (AEs) as well as follow-up for all AEs that have not been resolved will be recorded, changes to concomitant medications will be noted, vital signs will be taken, and efficacy evaluations will be performed as well. Investigators, site staff, subjects, and the study team will be blinded to the device assigned. The study includes collection of blood and urine samples. The end-of-treatment visit and the last estimation of glycemic control will occur at week 20 (visit 8) for all subjects. In addition, 2-week follow up will occur in order to collect safety data after the device is returned. The final visit will be at week 22 (visit 9). Subjects will be encouraged to complete all planned visits regardless of their adherence to study device administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 30 through 80 years;
2. Type 2 diabetes mellitus (T2DM) patients on stable oral anti-diabetic drugs for more than 3 months, and can maintain stable during study maintenance period;
3. HbA1c between 7.5 and 10% inclusive;
4. Subjects who are able and willing to perform self-monitoring of plasma glucose and self-administration of study device for the entire trial period;
5. Subjects who are able and willing to keep a diary;
6. Able and willing to sign informed consent and return for follow-up assessments.

Exclusion Criteria:

1. Subject has had any of the following new diagnoses within 1 year of screening:

   myocardial infarction, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure(NYHA III-IV), ventricular rhythm disturbances or thromboembolic disease;
2. Subjects with prior pancreatitis;
3. Subjects with insulin therapy (except for short term uses no longer than 7 days) or injectable antihyperglycemic agents (AHAs) within 3 months;
4. Female with a positive pregnancy test, planning to become pregnant during screening, active treatment, or the follow up period, breastfeeding, or judged to be using inadequate contraceptive methods;
5. Subjects who underwent previous intra abdominal, GI tract surgery or a major abdominal trauma within 6 months prior to screening visit;
6. Subjects with other implanted electrical stimulation devices;
7. Subject has any unresolved adverse skin condition in the area of device placement;
8. ALT/AST greater than 3 x upper limit of the institution's normal range (ULN) and/or total bilirubin ≥ 2.0 x ULN, active liver disease (other than nonalcoholic hepatic steatosis), including chronic active hepatitis B or C, hepatic cirrhosis, primary biliary cirrhosis, or active symptomatic gallbladder disease;
9. Subjects with moderate or severe renal impairment (serum creatinine ≥1.5 mg/dL in males or ≥ 1.4 mg/dL in females or urine microalbumin-creatinine ratio (ACR) >300 mg/g), conditions of congenital renal glucosuria, unstable or rapid progressing renal disease;
10. Has blood dyscrasias or any disorders causing hemolysis or unstable red blood cells or any other clinically significant hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia, coagulopathy);
11. Subjects with acute metabolic complications (such as ketoacidosis, lactic acidosis or hyperosmolar), proliferative diabetic retinopathy or macular edema within 6 months before screening;
12. Subjects with a history of malignancy ≤5 years prior to screening, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer;
13. Subjects a history of alcohol or drug abuse within 1 year prior to screening;
14. Subjects who received another investigational agent within 30 days prior to screening;
15. Subjects who are unlikely to be available for follow-up as specified in the protocol;
16. Subjects with a past or present psychiatric condition that may impair his or her ability to comply with the study procedures;
17. Subjects with conditions that, in the judgment of the investigator, precludes successful participation to the study;
18. Subjects with fever(body temperature> 37.5°C), perceptual function lost, or any metal implants.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c values to evaluate of the effect of DW1330 | 24 weeks, 2 weeks of screening, 20 weeks of treatment, and 2 weeks of post-treatment follow-up
  The primary study objective is to demonstrate the use of DW1330 is associated with improvement of blood glucose control, as measured by changes in glycated hemoglobin (HbA1c) values in comparison with placebo on blood glucose control parameters after 20 weeks of treatment. The time frame includes 2 weeks of screening, 20 weeks of treatment, and 2 weeks of post-treatment follow-up.

SECONDARY OUTCOMES:
To evaluate the change from baseline in the percentage of subject who achieve HbA1c < 7% | 24 weeks, 2 weeks of screening, and 20 weeks of treatment
  compare the test group and placebo group in percentage of subjects who achieve HbA1c < 7%
Change from baseline in FPG | baseline at visit 2, and visit 3, 4, 5, 6, 7, 8 of treatment [up to 20 weeks]
  Change from baseline in Fasting plasma glucose compare with test and control group
Evaluate the efficacy of SMBG | baseline at visit 2, and visit 4, 6, 8 of treatment [up to 20 weeks]
  Change from baseline in evaluate the efficacy of self monitoring blood glucose
Change from baseline in body weight | baseline at visit 2, and visit 3, 4, 5, 6, 7, 8 of treatment [up to 20 weeks]
  Change from baseline in body weight compare with test and control group
Change from baseline in OAD drugs description | baseline at visit 2, and visit 3, 4, 5, 6, 7, 8 of treatment [up to 20 weeks]
  compare the change of OAD drugs description following a 20 weeks treatment of DW1330 versus placebo

OTHER OUTCOMES:
Change from baseline of inflammatory biomarkers | baseline at 2 week,and 20 week
  The exploratory objective is to detect the change of biomarkers related to body glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Ming Chuang, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (6):
- Taiwan (6):
  - Chia-Yi Christian Hospital, Chiayi City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided